CLINICAL TRIAL: NCT06339827
Title: ASk Questions in GYnecologic Oncology (ASQ-GYO): A Randomized Controlled Trial of a Question Prompt List Communication Intervention in Outpatient Gynecologic Oncology Clinics
Brief Title: ASk Questions in GYnecologic Oncology (ASQ-GYO)
Acronym: ASQ-GYO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ira Winer (Other)
Responsible Party: Sponsor-Investigator, Ira Winer, Principle Investigator, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-102
Record Dates: First submitted 2024-03-21; First posted 2024-04-01 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Cervical Cancer; Vulvar Cancer; Vaginal Cancer; Gestational Trophoblastic Disease
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Gestational Trophoblastic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of the ASk Questions in GYnecologic Oncology (ASQ-GYO) Question Prompt List (Experimental): Participants are provided with a question prompt list
  Interventions: Behavioral: Administration of the ASk Questions in GYnecologic Oncology (ASQ-GYO) Question Prompt List
- No administration of the ASk Questions in GYnecologic Oncology (ASQ-GYO) Question Prompt List (No Intervention): Participants will not be provided with the question prompt list

INTERVENTIONS:
Behavioral: Administration of the ASk Questions in GYnecologic Oncology (ASQ-GYO) Question Prompt List — Participants are randomized and will receive the ASQ-GYO prompt list within 2 weeks prior to their new patient appointment with the gynecology oncology physician.
  Arms: Administration of the ASk Questions in GYnecologic Oncology (ASQ-GYO) Question Prompt List

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of the ASk Questions in GYnecologic Oncology question prompt list (ASQ-GYO QPL) at improving patient self-efficacy, distress, physician trust, and knowledge compared to usual care during new patient gynecologic oncology visits. Also to determine the acceptability of the ASQ-GYO QPL with new gynecologic oncology patients.

DETAILED DESCRIPTION:
* Potential participants who are scheduled for a new patient appointment will be contacted via phone or email to determine if they are interested in participating.
* If a participant is interested, they will choose their preferred method of consenting (phone, email, or in person) and if they would like to complete the pre-visit survey now or at a later time prior to their appointment
* If consented, all participants will be provided with the pre-survey questionnaire. If eligible, participants will then be randomized to usual care or the intervention (ASk Questions in GYnecologic Oncology question prompt list (ASQ-GYO QPL)
* If randomized to receive the ASQ-QYO QPL, they will be emailed this document and given a paper copy of the ASQ-GYO QPL in the waiting room prior to their visit to ensure they have received the intervention.
* Directly after the participant's visit, all participants will be asked to complete the post-visit survey on a tablet in the clinic waiting room, or via a secure link in an email within 1 week of the appointment.
* After completion of the post-visit survey and within one month of their visit, participants who were not randomized to receive the ASQ-GYO QPL will be sent the ASQ-GYO QPL via email so that they may also have access to this resource.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Understands spoken and written English
* Able to consent to study participation
* Biopsy confirmed gynecologic cancer diagnosis (ovarian, endometrial, cervical, vulvar, or vaginal cancer or Gestational Trophoblastic Disease) OR have imaging and/or laboratory findings highly concerning for a cancer diagnosis and have not seen a Gynecologic Oncologist

Exclusion Criteria:

* pathologic diagnosis of dysplasia only (cervical, vulvar, or endometrial)
* History and/or imaging/laboratory findings more indicative of a non-cancer diagnosis
* Previous treatment discussion with a Gynecologic Oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in pre- and post-visit self-efficacy scores and compared by trial group | All participants will complete the PEPPI instrument twice: within 2 weeks of their first visit and again within 1 week after the visit.
  The Perceived Efficacy in Patient-Provider Interactions (PEPPI) instrument is a validated, 20-item, 5-point Likert scale tool designed to measure patient's self-efficacy in obtaining medical information and attention to their medical concerns from physicians.

SECONDARY OUTCOMES:
Change in pre- and post-visit National Comprehensive Cancer Network (NCCN) Distress Thermometer scores compared by trial group | All participants, Twice: within 2 weeks of the first visit and again within 1 week after the visit
  The NCCN Distress Thermometer is a one-question, 11-point Likert scale for patient-reported distress in the past week including today
Change in pre- and post-visit Trust in a Physician scores compared by trial group | All participants, Twice: within 2 weeks of the first visit and again within 1 week after the visit
  The Trust in a Physician score is a validated, 5-point Likert scale with higher scores indicating more trust. The metric addresses generic physician trust prior to the visit, and trust in the specific physician the patient saw during their visit for after the visit
Knowledge Screen | All participants will complete a post-visit knowledge screen once within 1 week after their visit
  The Knowledge Screen is a 10-item, 5-point Likert scale, investigator-developed set of questions designed to elicit understanding of the contents of the Question Prompt List with higher scores indicating more understanding.
Patient perceptions of the Question Prompt List | The patients in the intervention group will complete this within 1 week after their visit.
  This is a 15-item investigator-developed set of questions with 7 items utilizing a 5-point Likert scale and 8 items utilizing binary yes/no questions designed to elicit the acceptability of the Question Prompt List among the patients in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Winer, MD PhD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States